CLINICAL TRIAL: NCT00856154
Title: Vaccination With Autologous Dendritic Cells Pulsed With HIV-Antigens for Treatment of Patients With Chronic HIV-Infection. Phase I Trial
Brief Title: Vaccination With Autologous Dendritic Cells Pulsed With HIV-Antigens for Treatment of Patients With Chronic HIV-Infection
Acronym: HIVDCVac
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Collaborators: Hvidovre University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Gitte Kronborg / MD DMSc Chief Medical Doctor, Infectious Disease Department, University Hospital Hvidovre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT2006-000102-22; EudraCT 2006-000102-22
Record Dates: First submitted 2009-03-03; First posted 2009-03-05 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-03

CONDITIONS: HIV Infections
Keywords: HIV-1; HLA-A2; Therapeutic; Vaccine; treatment vaccine; treatment naive
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Peptides on autologous Dendritic Cells — 10 Peptides Pulsed onto 10e7 autologous macrophage-derived maturated dendritic cells administered s.c. week 0, 2, 4, 8.
  1. Gag150 RLLNAWVKV
  2. Gag433 FLGKIWPV
  3. Env 67 NIWATHACV
  4. Pol606 KLGKAGYVV
  5. Vpu66 ALVEMGHHV
  6. Vif101 GLADQLIHL
  7. Vif23 SLVKHHMYV
  8. Gag298 KRWIILGLNKIVRMY
  9. gp41 VWGIKQLQARVLAVERYLKD
  10. Padre AKXVAAWTLKAAA
  Other Names: Dendritic Cells; HIV-1 Peptides

SUMMARY:
Phase I test of concept study: In an attempt to induce new immunity to HIV-1 during untreated HIV-1 infection the investigators have identified relatively immune silent immune subdominant HLA-A2-restricted HIV-1 CTL epitopes that fit individuals with the HLA-A2 tissue type (about 50% of peoples in Denmark). Immunising with these conserved epitopes could induce new immunity and lower viral load so the patient will live longer before AIDS or Antiviral medicine and a lower viral load will limit spread in the population. As adjuvants the investigators used patients' own autologous Dendritic Cells generated from blood cells in vitro. 12 healthy male HIV-1 infected not in therapy individuals were used for this therapeutic vaccination and tested for safety and induction of new cellular CD8 and CD4 T-cell immunity.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive male
* Viral load >1000/ml
* CD4 count >300
* HLA-A2 tissue type
* 18-50 years of age
* Able to follow the instructions
* Informed consent

Exclusion Criteria:

* Treated with other experimental vaccines or immune modulatig medicine
* Other chronic infectious diseases
* Allergy or autoimmune disease

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2008-04 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety: no changes in the blood Hemoglobin, leucocytes, trombocytes, serum sodium,potassium,creatinine,phosphatase, ALAT,ASAT, bilirubin,CRP. No dose limiting toxicity defined as unwanted events defined by CTC version 3 definition as greade 3 or more. | 12 months

SECONDARY OUTCOMES:
Cellular Immunity induction | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anders Fomsgaard, MD DMSc, Study Chair — Statens Serum Institut
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Thorn M, Tang S, Therrien D, Kloverpris H, Vinner L, Kronborg G, Gerstoft J, Corbet S, Fomsgaard A. Sequence conservation of subdominant HLA-A2-binding CTL epitopes in HIV-1 clinical isolates and CD8+ T-lymphocyte cross-recognition may explain the immune reaction in infected individuals. APMIS. 2007 Jun;115(6):757-68. doi: 10.1111/j.1600-0463.2007.apm_595.x. PMID 17550385
- See also: Danish Medicines Agency — http://www.laegemiddelstyrelsen.dk
- See also: Danish register of persons in projects — http://www.datatilsynet.dk
- See also: Statens Serum Institut in Denmark (government institution) — http://www.ssi.dk